CLINICAL TRIAL: NCT03623646
Title: Cisplatin or ImmunoTHerapy in Association With Definitive Radiotherapy in HPV-related oropharyngEal Squamous Cell Carcinoma: a Randomized Phase II Trial.
Acronym: CITHARE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18 VADS 06
Record Dates: First submitted 2018-08-02; First posted 2018-08-09 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma
Keywords: Oropharyngeal Squamous Cell Carcinoma; Anti PD-L1; Durvalumab; Radiation therapy; Cisplatin; Human Papilloma Virus
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (standard arm): Chemoradiotherapy arm (Other)
  Interventions: Drug: Chemoradiotherapy arm
- Arm B (Experimental arm): Immunotherapy + Radiotherapy arm (Experimental)
  Interventions: Drug: Immunotherapy + Radiotherapy arm

INTERVENTIONS:
Drug: Chemoradiotherapy arm — Radiation Therapy in combination with Chemotherapy (Cisplatin)
  Arms: Arm A (standard arm): Chemoradiotherapy arm
Drug: Immunotherapy + Radiotherapy arm — Radiation Therapy in combination with Immunotherapy drug (Durvalumab)
  Arms: Arm B (Experimental arm): Immunotherapy + Radiotherapy arm

SUMMARY:
This study is a phase II, multicenter, open-label study that has been designed to evaluate the efficacy and the safety of definitive Radiotherapy (RT) (70 Gy) delivered in combination with the anti-PD-L1 Durvalumab immunotherapy in patients with Human Papilloma Virus (HPV)-related oropharyngeal squamous cell carcinoma.

In this phase II trial, patients will be assigned in one of the two treatment arms:

* Arm A (standard arm): Chemoradiotherapy arm
* Arm B (Experimental arm): Immunotherapy + Radiotherapy arm

Total duration of treatment will be 6 months (at maximum in the experimental arm).

Patients will be followed for a maximum of 2 years following the date of randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, histologically proven squamous cell carcinoma of oropharynx T1 N1-N2 or T2-T3 N0 to N2 (AJCC 2018)
2. HPV positive status (positive staining for p16 in immunochemistry)
3. Presence of at least one measurable lesion according to RECIST v1.1 criteria (longest diameter recorded ≥10 mm with CT scan)
4. No prior anticancer therapy for OSCC
5. Patient eligible for definitive radiochemotherapy
6. Age ≥ 18 years
7. WHO performance status < 2 i.e. 0 or 1
8. Body weight >30kg
9. Life expectancy more than 3 months
10. Adequate Hematology laboratory data within 6 weeks prior to start of treatment: Absolute neutrophils> 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hemoglobin ≥ 9 g/dL
11. Adequate Biochemistry laboratory data within 6 weeks prior to start of treatment: Total bilirubin ≤ 1.5 x upper the normal limit, Transaminases ≤ 2.5 xUNL, Alkalin phosphatases ≤ 5 x UNL, Creatinin clearance ≥ 60 mL/min (Cockcroft), Glycemia ≤ 1.5 x UNL
12. Adequate Hemostasis laboratory data within 6 weeks prior to start of treatment: TP within the normal range
13. Women should be post-menopaused or willing to accept the use an effective contraceptive regimen during the treatment period and at least 3 months (durvalumab arm) or 6 months (cisplatin arm) after the end of the study treatment. All non-menopaused women should have a negative pregnancy test within 72 hours prior to registration. Men should accept to use an effective contraception during treatment period and at least 3 months (durvalumab arm) or 6 months (cisplatin arm) after the end of the study treatment
14. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
15. Signed written informed consent

Exclusion Criteria:

1. T1 N0, T1-T3 N3, T4 N0-N3, p16 + OSCC
2. Previous treatment with another check-point inhibitor
3. Other histologies : UCNT, p16- SCCHN, sino-nasal tumors
4. Patient ineligible for Cisplatin according to the updated SmPC of the drug (including patient with auditory deficiency, patient with neuropathy induced by previous Cisplatin treatment or patient treated with prophylactic phenytoin)
5. Metastatic disease
6. Previous radiotherapy, except anterior strictly out of field radiotherapy, received for treatment of another primary tumor considered in remission in the past 5 years
7. Participation in another therapeutic trial within the 30 days prior to entering this study
8. Uncontrolled disease such as diabetes, hypertension, symptomatic congestive heart or pulmonary failure, renal or hepatic chronic diseases... (non-exhaustive list)
9. Clinically significant cardiac disease or impaired cardiac function, such as:

   * Congestive heart failure requiring treatment (New York Heart Association (NYHA) Grade ≥ 2), left ventricular ejection fraction (LVEF) < 50% as determined by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO), or uncontrolled arterial hypertension defined by blood pressure > 140/100 mm Hg at rest (average of 3 consecutive readings),
   * History or current evidence of clinically significant cardiac arrhythmias, atrial fibrillation and/or conduction abnormality, e.g. congenital long QT syndrome, high- Grade/complete AV-blockage
   * Acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft (CABG), coronary angioplasty, or stenting), < 3 months prior to screening
   * QT interval adjusted according to Fredericia (QTcF) > 470 msec on screening ECG
10. Current or prior use of immunosuppressive medication within 28 days before the first fraction of RT (exception: systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or equivalent are allowed as well as steroids as premedication for hypersensitivity reactions (eg, CT scan premedication) - Topical, inhaled, nasal and ophthalmic steroids are not prohibited)
11. Active suspected or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, irritable bowel syndrome, Wegner's granulomatosis and Hashimoto's thyroiditis, diverticulitis with the exception of diverticulosis, systemic lupus erythematosus, Sarcoidosis syndrome). Note: participants with vitiligo or alopecia, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, patients with celiac disease controlled by diet alone, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger, are permitted to enroll
12. Known primary immunodeficiency or active HIV (positive HIV 1/2 antibodies)
13. Known active or chronic viral hepatitis or history of any type of hepatitis within the last 6 months indicated by positive test for hepatitis B surface antigen (HBV sAG) or hepatitis C virus ribonucleic acid (HCV antibody)
14. History of organ transplant requiring use of immunosuppressive medication
15. History of active tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice)
16. Current pneumonitis or interstitial lung disease
17. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
18. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease
19. History of severe allergic reactions to any unknown allergens or any components of the study drug
20. History of leptomeningeal carcinomatosis
21. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

    1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician
    2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician
22. Uncontrolled severe infectious disease, active hemorrhagic syndrome
23. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP
24. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
25. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP
26. Vaccination for yellow fever
27. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of cisplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
The rate of patients alive without progression at 12 months. | 12 months for each patient

SECONDARY OUTCOMES:
Progression-free survival. | 24 months for each patient
Overall survival. | 24 months for each patient
Safety will be evaluated using National Cancer Institute Common Toxicity Criteria Adverse Event (NCI-CTCAE) version 4.03. | 24 months for each patient
Quality of life will be evaluated using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30). | 24 months for each patient
Quality of life will be evaluated using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Head & Neck 35 (EORTC QLQ-H&N35). | 24 months for each patient

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Bordeaux, Bordeaux
  - Institut Universitaire du Cancer Toulouse (IUCT-O), Toulouse